CLINICAL TRIAL: NCT03418766
Title: The Relationship Between Right-to-left Shunt and Brain White Matter Lesions in Chinese Patients With Migraine:a Multicenter Study. CAMBRAIN Study.
Brief Title: The Relationship Between Right-to-left Shunt and Brain White Matter Lesions in Patients With Migraine
Acronym: CAMBRAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: CAMBRAIN
Record Dates: First submitted 2018-01-16; First posted 2018-02-01 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-03

CONDITIONS: White Matter Disease; Right-to-left Shunt; Migraine Disorders
Keywords: Right-to-left Shunt; Brain White Matter Lesions; Migraine
MeSH Terms: conditions — Leukoencephalopathies; Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal: Normal healthy individual without migraine.
- Magraine: Clinical history of migraine diagnosed by a neurologist according to the International Classification of Headache Disorders.

SUMMARY:
The purpose of the study is to evaluate the prevalence of white matter lesions in Chinese migraineurs with and without right-to-left shunt. The aim is to study the relationship among right-to-left shunt, migraine and white matter lesions.

DETAILED DESCRIPTION:
This is a prospective multicenter study of Chinese population. Participants (normal individuals without migraine and migraineurs) are included after standardized diagnostic procedures (TCD and migraine diagnosis). For all the participants, brain MRI and c-TCD are required. Up to 10-15 study sites nationwide will be needed to recruit the planned participant population during a 1-year period.

The information of each participants will be registered, including basic facts, the longitudinal headache history, frequency, location, quality, intensity, duration, accompanied symptoms, precipitating and exacerbating factors, with or without aura, and Headache Impact Test-6 (HIT-6) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients who fulfilled the criteria for migraine according to the International Classification of Headache Disorders III-beta were included.

healthy volunteers without a history of migraine were included as controls.

Exclusion Criteria:

* Subjects were excluded from the study if they had severe arterial stenosis, an insufficient temporal window, inadequate cubital venous access, and/or were unable to perform the Valsalva manoeuvre (VM) because of severe heart or lung disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We detect RLS through contrast-enhanced transcranial Doppler (c-TCD). The normal individuals will be selected to group 1, while those who suffer from migraine will be selected to group 2. All the participants are required to take c-TCD and brain MRI.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
contrast-enhanced transcranial Doppler (c-TCD) | 1 year
  Brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Yingqi Xing, MD,PhD, Study Chair — The First Hospital of Jilin University; Sibo Wang, MD,PhD, Principal Investigator — The First Hospital of Jilin University; Yi Yang, MD,PhD, Study Director — The First Hospital of Jilin University; Yongsheng Gao, MD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First hospital of Jilin Uni, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Del Sette M, Dinia L, Bonzano L, Roccatagliata L, Finocchi C, Parodi RC, Sivori G, Gandolfo C. White matter lesions in migraine and right-to-left shunt: a conventional and diffusion MRI study. Cephalalgia. 2008 Apr;28(4):376-82. doi: 10.1111/j.1468-2982.2008.01544.x. Epub 2008 Feb 22. PMID 18294247